CLINICAL TRIAL: NCT04607915
Title: Technology-enabled Collaborative Care for Diabetes (TECC-Diabetes) Management During COVID: A Feasibility Study
Brief Title: Technology-enabled Collaborative Care for Diabetes Management During COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Peter Selby, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 104-2020
Record Dates: First submitted 2020-07-30; First posted 2020-10-29 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention for TECC Model (Experimental)
  Interventions: Behavioral: Intervention for TECC Model

INTERVENTIONS:
Behavioral: Intervention for TECC Model — The Care Coordinator (CC) will provide brief coaching sessions (15 to 20 minutes) to each participant once per week for 8 weeks. Participants can identify topics for discussion and the CC and participant can decide if a video session via WebEx is required versus a phone call. Also, participants will be given peer support and will be indirectly monitored by a virtual care team of experts.

SUMMARY:
The overall goal of this research program is to evaluate the effectiveness of a Technology-Enabled Collaborative Care program. In this study, we examine the feasibility of such a program, called the Technology-Enabled Collaborative Care (TECC) for type 2 diabetes designed to support patients with diabetes and mental health concerns during COVID-19.

DETAILED DESCRIPTION:
There is growing concern regarding the impact of COVID-19 and social isolation on mental health and wellbeing, particularly adults living with type 2 diabetes (T2DM), who are at greater risk for mental health issues than the general population. Self-management education and support for healthy eating, physical activity, glucose monitoring, medication adherence and problem solving are vital components of diabetes care. Due to social distancing and limited care and resources, that are likely to persist in the post pandemic phase other innovative service models should be developed and adopted to improve service delivery. The overall goal of this research program is to evaluate the effectiveness of a Technology-Enabled Collaborative Care program. In this study, we examine the feasibility of such a program, called the Technology-Enabled Collaborative Care (TECC) for T2DM designed to support patients with diabetes and mental health concerns during COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and older
* Clinician diagnosis of Type 2 diabetes for at least one year
* A1C level of 7.5% or higher within the last 6 months (benchmark is 7%)
* Access to telephone or internet through computer or mobile
* Experiencing some distress, score of ** on Perceived Stress Scale

Exclusion Criteria:

* Unable to provide consent
* Unable to understand English
* Pregnant or planning to get pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment Numbers | Through the study completion, an average of 4 months
  The primary outcome in this study is feasibility, specifically process outcomes. This includes assessing recruitment number
Feasibility - Participant characteristics | up to 8-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes participant characteristics
Feasibility - Participant Engagement (retention rate) | up to 8-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes participant retention rate (e.g., defined by time between first and last visit)
Feasibility - Participant Engagement (intensity) | up to 8-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes intensity (e.g., number of session participants attend)
Feasibility - Participant Engagement (drop out) | up to 8-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes drop out (consented/enrolled but did not attend first one-on-one)
Feasibility - Delivery of Intervention (Time with coach) | up to 8-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes the amount of time a coach spends per interaction
Feasibility - Delivery of Intervention (Mode of interaction) | up to 12-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes the mode of the interaction (i.e., virtual, telephone or both)
Feasibility - Delivery of Intervention (Coach strategies) | up to 12-weeks
  The primary outcome in this study is feasibility, specifically process outcomes. This includes what strategies are used by the coach (i.e., educational, psychosocial support, behaviour modifications, or case management/monitoring)

SECONDARY OUTCOMES:
Study Participant experience and satisfaction via semi-structured interview | up to 8-weeks
  The secondary outcome consists of study participant experience/satisfaction.
Care Coordinator experience and satisfaction via semi-structured interview | up to 8-weeks
  The secondary outcome consists of Care Coordinator experience and satisfaction.
Virtual Care Team experience and satisfaction via semi-structured interview | up to 8-weeks
  The secondary outcome consists of Virtual Care Team experience and satisfaction.

OTHER OUTCOMES:
Exploratory Outcome - Health Behaviour metrics (physical activity) | up to 4-weeks
  The exploratory outcomes will include Health Behaviour metrics via International Physical Activity Questionnaire). Individual scores per question, the higher the score means the higher the level of physical activity.
Exploratory Outcome - Health Behaviour metrics (diet) | up to 4-weeks
  The exploratory outcomes will include Health Behaviour metrics (via Mediterranean Diet Adherence Screener Modified (MEDAS modified)
Exploratory Outcome - Health Behaviour metrics (confidence/importance to change behaviour) | up to 12-weeks
  The exploratory outcomes will include Health Behaviour metrics (via readiness to change ruler (smoking, alcohol, nutrition, physical activity). Minimum score: 0; maximum score: 10; higher score represented a better outcome.
Exploratory Outcome - Substance Use (GAINS-SS) | up to 12-weeks
  The exploratory outcomes will include substance use (via GAINS-SS (Global Appraisal of Individual Needs- Short Screener). Minimum score: 0; maximum score: 20; higher score represented a worse outcome.
Exploratory Outcome - Substance Use (alcohol) | up to 12-weeks
  The exploratory outcomes will include substance use (Alcohol Use Disorders Identification Test (AUDIT); Minimum score: 0; maximum score: 40; higher score represented a worse outcome.
Exploratory Outcome - Substance Use | up to 12-weeks
  The exploratory outcomes will include substance use (via heaviness of smoking index - 2 items out of Fagerstrom test for nicotine dependence (FTND)); Minimum score: 0; maximum score: 6; higher score represented a worse outcome.
Exploratory Outcome - Mental Health (depression) | up to 12-weeks
  The exploratory outcomes will include Mental Health measures (via Patient Health Questionnaire (PHQ-9)). Minimum score: 0; maximum score: 27; higher score represented a worse outcome.
Exploratory Outcome - Mental Health (Anxiety) | up to 12-weeks
  The exploratory outcomes will include Mental Health measures via Generalized Anxiety Disorder-7 (GAD-7). Minimum score: 0; maximum score: 21; higher score represented a worse outcome.
Exploratory Outcome - Mental Health (Diabetes awareness/insight) | up to 12-weeks
  The exploratory outcomes will include Mental Health measures via Diabetes awareness and insight scale. Minimum score: 0; maximum score: 10; higher score represented a better outcome.
Exploratory Outcome - Mental Health (Diabetes Distress) | up to 12-weeks
  The exploratory outcomes will include Mental Health measures via Diabetes Distress Scale. Minimum score: 0; maximum score: 6; higher score represented a worse outcome.
Exploratory Outcome - Mental Health (Stress) | up to 12-weeks
  The exploratory outcomes will include Mental Health measures via perceived stress scale (PSS). Minimum score: 0; maximum score: 40; higher score represented a worse outcome (i.e., higher perceived stress).
Exploratory Outcome - Quality of Life | up to 12-weeks
  The exploratory outcomes will include quality of life (via European Quality of Life - 5 Dimensions scale - EQ5D). Minimum score: 0; maximum score: 100; higher score represented a better outcome.
Exploratory Outcome - Quality of Life | up to 12-weeks
  The exploratory outcomes will include quality of life (via Verona satisfaction scale). Minimum score: 0; higher score represented a better outcome.
Exploratory Outcome - Waist circumference | up to 12-weeks
  self-report
Exploratory Outcome - BMI (height/weight) | up to 12-weeks
  self-report
Exploratory Outcome - Blood pressure | up to 12-weeks
  self-report
Exploratory Outcome - Current medication | up to 12-weeks
  list
Exploratory Outcome - Blood work | up to 12-weeks
  Hemoglobin A1C levels
Exploratory Outcome - Pain | up to 12-weeks
  Brief Pain Inventory-sf. Minimum score: 0; maximum score: 10; higher score represented a worse outcome (i.e., more pain).
Exploratory Outcome - Diabetes duration | up to 12-weeks
  months
Exploratory Outcome - Diabetes self-management | up to 12-weeks
  Diabetes Self-Management and Technology Questionnaire (DSMT-Q); Minimum score: 0; maximum score: 48; higher score represented a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Selby, Principal Investigator — CAMH; Diana Sherifali, Principal Investigator — McMaster University; Farooq Naeem, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Vojtila L, Sherifali D, Dragonetti R, Ashfaq I, Veldhuizen S, Naeem F, Agarwal SM, Melamed OC, Crawford A, Gerretsen P, Hahn M, Hill S, Kidd S, Mulsant B, Serhal E, Tackaberry-Giddens L, Whitmore C, Marttila J, Tang F, Ramdass S, Lourido G, Sockalingam S, Selby P. Technology-Enabled Collaborative Care for Concurrent Diabetes and Distress Management During the COVID-19 Pandemic: Protocol for a Mixed Methods Feasibility Study. JMIR Res Protoc. 2023 Jan 17;12:e39724. doi: 10.2196/39724. PMID 36649068